CLINICAL TRIAL: NCT06999850
Title: Implementazione e Validazione di un Test Per l'Analisi Del Movimento Della Salita e Discesa Delle Scale Con Sensori Indossabili
Brief Title: Implementation and Validation of Instrumented Stair Climb Test
Acronym: SCTS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Politecnico di Milano (Other); ASP Istituti Milanesi Martinitt e Stelline e Pio Albergo Trivulzio (Unknown); Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: 106_24 (ex1134)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Stair Climbing; Instrumentation; Test
Keywords: Stair Climb Test; Cerebral Palsy; Stroke; amputee; Parkinson
MeSH Terms: conditions — Cerebral Palsy; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- healthy children: This group involves healthy children aged 4-18 years old, without gait impairmets
  Interventions: Other: Walk Test; Other: Repaeted Instrumented Stair Climb Test
- Healthy adults: This group involves healthy adults aged 18-65 years old, without gait impairmets
  Interventions: Other: Walk Test; Other: Repaeted Instrumented Stair Climb Test
- Healthy elderly: This group involves healthy eleferly aged 65-85 years old, without gait impairmets
  Interventions: Other: Walk Test; Other: Repaeted Instrumented Stair Climb Test
- CP subjects: pediatric subjects diagnosed with Infantile Cerebral Paralysis (PCI) and clinical sign of left or right hemiparesis;
  Interventions: Other: Instrumented Stair Climb Test; Other: Walk Test
- Leg amputee subjects: Patients aged 19-80 years, with results of leg amputation (transtibial), who carry limb prostheses
  Interventions: Other: Instrumented Stair Climb Test; Other: Walk Test
- Arthroplasty Subjects: patients aged 65-80 years, with aftereffects of hip or knee arthroplasty, excluding prosthetic revision procedures
  Interventions: Other: Instrumented Stair Climb Test; Other: Walk Test
- Parkinson Subjects: atients aged 65-80 years, with diagnosis of Parkinson's disease or Parkinsonism even on a vascular basis
  Interventions: Other: Instrumented Stair Climb Test; Other: Walk Test
- Stroke Subjects: Patients aged 65-80 years, with aftereffects of Cerebral Stroke with left or right hemiparesis
  Interventions: Other: Instrumented Stair Climb Test; Other: Walk Test

INTERVENTIONS:
Other: Instrumented Stair Climb Test — Instrumented test of climbing and descending stairs for the evaluation of kinematic and electromyographic variables. The test consists of repeating the ascent and descent of a flight of 10-12 steps;
  Groups: Arthroplasty Subjects; CP subjects; Leg amputee subjects; Parkinson Subjects; Stroke Subjects
Other: Walk Test — Assessment of climbing and walking skills through test series:
  Borg scale: An evaluation scale for measuring effort perception. The evaluation scale consists of answering some questions at the end of the exercise described above; 10-metre walk test (10MWT): Test to assess walking speed in metres per second over a short distance. Can be used to determine functional mobility, gait and vestibular function. The test consists of walking at a steady speed and safely for 10 metres; 30 second sit to stand test: test for the evaluation of strength and endurance of the legs in the elderly. The test consists in performing the movement of standing up and sitting down from a chair for 30 consecutive seconds; Timed Up & Go test (TUG): test to assess the risk of falling and balance. During the test, patients wear normal footwear and may use a walking aid if necessary. The patient starts in a sitting position, gets up on the therapist's command, walks in a straight line for a distance of 3 m
Other: Repaeted Instrumented Stair Climb Test — Instrumented test of climbing and descending stairs for the evaluation of kinematic and electromyographic variables. The test consists of repeating the ascent and descent of a flight of 10-12 steps. In this case, the ascent and descent of the stairs must be repeated two times. Between the two trial the IMU units must be repositioned.
  Groups: Healthy adults; Healthy elderly; healthy children

SUMMARY:
The aim of this study is to design an instrumented test for the evaluation of the climb of stairs. In particular, the main purpose is to characterize and compare the performance of subjects, both pediatrics and adults, with different pathologies (cerebral palsy, amputee, Parkinson's disease, stroke and arthroplasty) in carrying out the instrumented test of climbing and descending stairs. This would provide potentially useful information to complement the clinical assessment, including investigating the existence of correlations between the instrumental data obtained and the clinical scales collected. The secondary objective is to evaluate, in a first phase of the study, the feasibility and reliability of the test, analyzing the validity of the indices obtained in terms of intra- and inter-operator reliability on healthy subjects.

DETAILED DESCRIPTION:
In today's clinical practice there are several assessment tools available to measure strength, endurance and balance. These tools include manual testing, standardised measurement scales or disease-specific scoring systems in which the results obtained during the performance of different motor tasks are calculated to obtain an overall score reflecting the functional level. Among the most used tests, for example, we remember the Six Minute Walking Test, in which the maximum distance walked, expressed in meters, is measured in a time of 6 minutes under standardized conditions, allowing the evaluation of muscular endurance and gait aspects. In addition to tests that monitor walking abilities, there are tests for more complex activities such as climbing and descending stairs. The ability to climb stairs, in contrast to flat walking, can be considered a more challenging task, as it places greater emphasis on muscle strength of lower limbs, requires a greater range of motion of the lower limb joints and increases the demand for posture control and balance system. In addition, falls from stairs can cause more serious injury or even death than falls on a floor. Therefore, for patients with a higher risk of falling, an objective assessment of the performance of climbing stairs could be of great interest, providing fundamental support in managing the activities of the patient's daily life. In the past, a number of methods and technologies have been proposed to analyse and quantify human gait. Measurement systems range from optoelectronic systems, pressure pads or force plates to mobile sensors worn on the body such as inertial units (IMUs) or pressure pads. Mobile gait analysis systems based on IMU, in particular, are attracting increasing interest for use in long-term assessments that can be easily performed in clinical practice. Similarly, inertial sensors could be adopted for an objective evaluation of the ascent and descent of ladders thanks to adapted step analysis algorithms capable of segmenting, parameterizing and classifying the ascent and descent of ladders. The aim of this study, therefore, is to design a test for the evaluation of climbing stairs based on the use of wearable sensors. In particular, the main objective will be to characterise and compare the performance of subjects with different pathologies, providing potentially useful information to complement clinical evaluation. The secondary objective of the study will be to analyse the reliability of the indices obtained. This work proposal is the result of collaboration between several centres: IRCCS E. Medea, IRCCS Istituti Clinici Maugeri Tradate, Pio Albergo Trivulzio and Politecnico di Milano. In particular, IRCCS E. Medea, IRCCS Istituti Clinici Maugeri Tradate and Pio Albergo Trivulzio will be responsible for the recruitment of subjects and data collection. These centres will have the support of the Politecnico di Milano for the processing of data and for the development of the algorithms necessary for the extraction of the monitored parameters from the devices used.

ELIGIBILITY:
Common inclusion criteria for all groups:

- Ability to climb and descend 10 steps with supervision, even with handrail support.

Common exclusion criteria for all groups:

* Need for help from an operator or use of orthoses to make the stairs;
* Inability to dress the instrumentation (accelerometer/electromyograph);
* clinical condition that does not recommend the execution of scales (e.g. NYHA Class IV cardiovascular decompensation, epilepsy not controlled by drugs, serious visual disturbances...);
* inability to follow verbal instructions.

Inclusion criteria for the healthy group :

* age 4-80 years (8 subjects 4-18 years; 8 subjects 19-65 years; 8 subjects 65-80 years);
* absence of diagnosis of neurological or orthopaedic pathologies, which impair the patient's mobility.

Inclusion criteria for the PCI group :

* age range 4-18 years;
* Diagnosis of Infantile Cerebral Palsy;
* right or left hemiparesis;
* ability motor skills in levels I - III according to the GMFCS (Gross Motor Function Classification System).

Inclusion criteria for the Orthopaedic group:

* Age 65-80 years;
* postoperative postoperative hip or knee arthroplasty (in election and post-fracture, any revisions will be excluded).

Inclusion criteria for the Amputee group:

* age range from 19 to 80 years;
* Leg amputation (trans-tibial), fitted with limb prosthesis.

Inclusion criteria for the Parkinson's group:

* age range from 65 years;
* diagnosis of Parkinson's disease or Parkinsonism also on a vascular basis.

Inclusion criteria for the group Ictus Cerebri:

* Age 65-80 years;
* Aftereffects of Ictus Cerebri;
* left or right hemiparesis.

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In the first validation phase of this project, healthy subjects will be involved, particularly a group of 8 subjects aged 4-18, a group of 8 subjects aged 19-65, and a group of 8 subjects aged 65-80.
  In the second phase of the project, patients belonging to 5 different groups will be involved: patients with Infantile Cerebral Palsy (PCI group), patients with postoperative aftereffects of hip or knee arthroplasty (orthopedic group), leg amputees (Amputee group), patients with Parkinson's disease (Parkinson group), and patients with Cerebral Stroke (Stroke group).
  64 participants will be enrolled in total for the study.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2026-04-04 (Estimated)

PRIMARY OUTCOMES:
Absolue error automatic test time | Through study completion, an average of 1 year
  Absolute errors were calculated for the duration time of the stair ascent and descent and for each variable by taking the absolute value after subtracting the values obtained using IMU methods from the value measured using the tradional chronometer method
Intra - inter operator variability | Through study completion, an average of 1 year
  To ensure consistency between the data obtained by the IMU method and the data obtained by the traditional chronometric method, the investigators first calculated the normality of the data. The two-way mixed effects model, absolute agreement, and average measurements were used to calculate the ICCs between the duration time of both systems in case of normality. Instead, the Sperman test was used by the investigator if the data had a non-normal distribution

SECONDARY OUTCOMES:
correlations with Ten meters Walk Test (10mWT) | Through study completion, an average of 1 year
  The investigators determine if there are any correlations between the instrumental data gathered from a test performed using the IMU method and the clinical test of the Ten meters walking test (10mWT). In the 10mWT the total time taken to ambulate 6 meters (m) is recorded to the nearest hundredth of a second. 6 m is then divided by the total time (in seconds) taken to ambulate and recorded in m/s.
correlations with 30 seconds chair to stand test | Through study completion, an average of 1 year
  The investigators determine if there are any correlations between the instrumental data gathered from a test performed using the IMU method and the clinical test of the 30 seconds chair to stand test. The test score is the total number of lifts completed in 30 seconds. During the test, the participant can stop and rest if he is tired without stopping time. If a person fails to perform any high the score for the test is zero
correlations with Timed Up and Go (TUG) | Through study completion, an average of 1 year
  The investigators determine if there are any correlations between the instrumental data gathered from a test performed using the IMU method and the clinical test Timed Up and Go test (TuG). The score in the text corresponds to the time taken by the participants to get up, walk to a distance of 3 m, turn around and return to their seats. Regular walking aids are permitted and recorded if necessary.
correlations with Borg Scale | Through study completion, an average of 1 year
  The investigators determine if there are any correlations between the instrumental data gathered from a test performed using the IMU method and the clinical Borg Scale. This is a scale to assess the intensity of exercise without having to rely on physiological parameters. The original Borg version is a scale of 6-20.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy